CLINICAL TRIAL: NCT03179904
Title: Phase II Trial to Evaluate the Efficacy of the FASN Inhibitor, TVB-2640, in Combination With Trastuzumab Plus Paclitaxel or Endocrine Therapy in Patients With HER2+ Metastatic Breast Cancer Resistant to Trastuzumab-Based Therapy
Brief Title: TVB-2640 and Trastuzumab With Paclitaxel or Endocrine Therapy for Treatment of HER2 Positive Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1633; W81XWH-16-1-0269 (Other Grant/Funding Number: Department of Defense); W81XWH-16-1-0268 (Other Grant/Funding Number: Department of Defense); NCI-2017-00944 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16-010066 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2017-05-30; First posted 2017-06-07 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Advanced Breast Carcinoma; HER2-Positive Breast Carcinoma; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; HER2-positive Breast Cancer
MeSH Terms: interventions — Anastrozole; TVB-2640; exemestane; Fulvestrant; Letrozole; Paclitaxel; Taxes; Trastuzumab; CT-P6; PF-05280014; Disulfides; Ogivri; Ontruzant; trastuzumab biosimilar HLX02; Magnetic Resonance Spectroscopy; X-Rays; Specimen Handling; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (FASN inhibitor TVB-2640, paclitaxel, trastuzumab) (Experimental): Patients receive FASN inhibitor TVB-2640 PO QD on days 1-28, paclitaxel IV over 1-96 hours on days 1, 8, and 15, and trastuzumab IV over 30-90 minutes on days 1, 8, 15, and 22 and optionally every 21 days after 3 cycles and paclitaxel is discontinued. Cycles repeat every 28 days in the absence of disease progression or unexpected toxicity. Patients also undergo ECHO and CT or MRI at screening and on study and undergo collection of blood samples and biopsy on study.
  Interventions: Drug: Denifanstat; Procedure: Echocardiography; Drug: Paclitaxel; Biological: Trastuzumab; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection; Procedure: Biopsy
- Cohort B (TVB-2640, trastuzumab, endocrine therapy) (Experimental): Patients receive FASN inhibitor TVB-2640 PO QD on days 1-28 and trastuzumab IV over 30-90 minutes on days 1, 8, 15, and 22 and optionally every 21 days after 3 cycles and paclitaxel is discontinued. Patients also continue endocrine therapy of either anastrozole PO QD, exemestane PO QD, fulvestrant IM on days 1 and 14 of cycle 1 and day 1 of subsequent cycles, or letrozole PO QD. Cycles repeat every 28 days in the absence of disease progression or unexpected toxicity. Patients also undergo ECHO and CT or MRI at screening and on study and undergo collection of blood samples and biopsy on study.
  Interventions: Drug: Anastrozole; Drug: Denifanstat; Drug: Exemestane; Drug: Fulvestrant; Procedure: Echocardiography; Drug: Letrozole; Biological: Trastuzumab; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection; Procedure: Biopsy

INTERVENTIONS:
Drug: Anastrozole — Given PO
  Other Names: Anastrazole; Arimidex; ICI D1033; ICI-D1033; ZD-1033
  Arms: Cohort B (TVB-2640, trastuzumab, endocrine therapy)
Drug: Denifanstat — Given PO
  Other Names: ASC 40; ASC-40; ASC40; FASN Inhibitor TVB-2640; TVB 2640; TVB-2640; TVB2640
Drug: Exemestane — Given PO
  Other Names: Aromasin; FCE-24304
  Arms: Cohort B (TVB-2640, trastuzumab, endocrine therapy)
Drug: Fulvestrant — Given IM
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ZD9238
  Arms: Cohort B (TVB-2640, trastuzumab, endocrine therapy)
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara
  Arms: Cohort B (TVB-2640, trastuzumab, endocrine therapy)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Cohort A (FASN inhibitor TVB-2640, paclitaxel, trastuzumab)
Biological: Trastuzumab — Given IV
  Other Names: 180288-69-1; ABP 980; ALT02; Biceltis; CANMab; CT-P06; CT-P6; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Herclon; Hertraz; Herzuma; Immunoglobulin G 1 (Human-Mouse Monoclonal RhuMab HER2gamma1-Chain Antihuman p185(Sup c-erbB2) Receptor); Disulfide with Human-Mouse Monoclonal RhuMab HER2 Light Chain; Dimer; Kanjinti; Ogivri; Ontruzant; PF-05280014; QL 1701; QL-1701; QL1701; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; Trastuzumab Biosimilar CT-P6; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar QL1701; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-pkrb; Trastuzumab-qyyp; Trazimera
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT SCAN; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI; Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI Scan; MRIs; NMRI; nuclear magnetic resonance imaging; sMRI; Structural MRI
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx

SUMMARY:
This phase II trial studies how well FASN inhibitor TVB-2640, paclitaxel, and trastuzumab work in treating patients with HER2 positive breast cancer that has spread to other places in the body (metastatic). FASN inhibitor TVB-2640 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Trastuzumab is a form of targeted therapy because it attaches itself to specific molecules (receptors) on the surface of cancer cells, known as HER2 receptors. When trastuzumab attaches to HER2 receptors, the signals that tell the cells to grow are blocked and the cancer cell may be marked for destruction by the body's immune system. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Estrogen can cause the growth of breast cancer cells. Drugs used in endocrine therapy either lower the amount of estrogen made by the body or blocks the use of estrogen by the tumor cells. This may help stop the growth of tumor cells that need estrogen to grow. Giving FASN inhibitor TVB-2640 and trastuzumab in combination with paclitaxel or endocrine therapy may help control the disease in patients with HER2 positive breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the overall tumor response rate (ORR i.e. complete response [CR]+partial response [PR]) of the combination of FASN inhibitor TVB-2640 [TVB-2640] with paclitaxel and trastuzumab in patients with taxane and trastuzumab-resistant, advanced HER2-positive breast cancer.

II. To estimate the ORR of the combination of TVB-2640 with paclitaxel and trastuzumab in patients with taxane and trastuzumab-resistant, advanced HER2-positive breast cancer.

SECONDARY OBJECTIVES:

I. For each patient cohort, to evaluate the safety profile of the combination of TVB-2640 with paclitaxel and trastuzumab.

II. For each patient cohort, to assess the clinical benefit rate (CBR), duration of response, and progression free survival of the combination of TVB-2640 with paclitaxel and trastuzumab.

III. To obtain a point and interval estimate of the difference in RR as well as the difference in CBR between cohort A and cohort B.

CORRELATIVE RESEARCH OBJECTIVES:

I. For each patient cohort, to assess the changes in FASN, phosphorylation (p)AKT, and pS6 expression in tumor tissue after the first cycle of the combination of TVB-2640 with paclitaxel and trastuzumab from pre-treatment levels.

II. For each patient cohort, to assess the changes in levels of cellular apoptosis in tumor tissue after the first cycle of the combination of TVB-2640 with paclitaxel and trastuzumab from pre-treatment levels.

III. For each patient cohort, to assess the changes in serum FASN after the first cycle of the combination of TVB-2640 with paclitaxel and trastuzumab from pre-treatment levels.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT A: Patients receive FASN inhibitor TVB-2640 orally (PO) once daily (QD) on days 1-28, paclitaxel intravenously (IV) over 1-96 hours on days 1, 8, and 15, and trastuzumab IV over 30-90 minutes on days 1, 8, 15, and 22, and optionally every 21 days after 3 cycles and paclitaxel is discontinued. Cycles repeat every 28 days in the absence of disease progression or unexpected toxicity. Patients also undergo echocardiography (ECHO) and computed tomography (CT) or magnetic resonance imaging (MRI) at screening and on study and undergo collection of blood samples and biopsy on study.

COHORT B: Patients receive FASN inhibitor TVB-2640 PO QD on days 1-28 and trastuzumab IV over 30-90 minutes on days 1, 8, 15, and 22 and optionally every 21 days after 3 cycles and paclitaxel is discontinued. Patients also continue endocrine therapy of either anastrozole PO QD, exemestane PO QD, fulvestrant intramuscularly (IM) on days 1 and 14 of cycle 1 and day 1 of subsequent cycles, or letrozole PO QD. Cycles repeat every 28 days in the absence of disease progression or unexpected toxicity. Patients also undergo ECHO and CT or MRI at screening and on study and undergo collection of blood samples and biopsy on study.

After completion of study treatment, patients are followed up every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION INCLUSION CRITERIA
* Age >=18 years
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria that is:

  * A non-nodal lesion is considered measurable if its longest diameter can be accurately measured as >= 1.0 cm with computed tomography (CT) scan, CT component of a positron emission tomography (PET)/CT, or magnetic resonance imaging (MRI) and/or
  * A malignant lymph node is considered measurable if its short axis is > 1.5 cm when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm)
  * Note: tumor lesions in a previously irradiated area are not considered measurable disease; disease that is measurable by physical examination only is not eligible
* Received =< six (6) prior chemotherapy regimens in the metastatic setting
* Cohort A one of the following must be true:

  * Distant disease progression during administration of combination therapy with taxane based chemotherapy and anti-HER2 therapy (trastuzumab or pertuzumab) for metastatic disease

    * Note: patients who began treatment with this combination and discontinued taxane-based chemotherapy due to intolerability before distant disease progression are eligible
  * Distant disease progression during administration or within 180 days of discontinuing combination therapy with taxane based chemotherapy and anti-HER2 therapy (trastuzumab or pertuzumab) in the adjuvant disease

    * Note: patients who began treatment with this combination and discontinued taxane-based chemotherapy due to intolerability before distant disease progression are eligible
  * For patient who received taxane based chemotherapy and anti-HER2 therapy (trastuzumab or pertuzumab) in the neo-adjuvant setting and underwent surgical resection of primary breast disease: distant disease progression during or within 180 days of discontinuing anti-HER2 therapy (trastuzumab or pertuzumab) in the adjuvant setting
* Cohort B (one of the following must be true):

  * Distant disease progression during administration of combination therapy with endocrine therapy and anti-HER2 therapy (trastuzumab or pertuzumab) for metastatic disease; permissible endocrine therapies include an aromatase inhibitor or fulvestrant

    * NOTE: Tamoxifen is not permissible
  * Distant disease progression during administration of combination therapy with endocrine therapy and anti-HER2 therapy (trastuzumab or pertuzumab) in the adjuvant setting; permissible endocrine therapies include an aromatase inhibitor or fulvestrant

    * NOTE: Tamoxifen is not permissible
* Willingness to provide mandatory tumor tissue specimens for correlative research

  * NOTE: If insufficient or no tissue is obtained by the pre-registration biopsy, an archival tissue specimen (preferably from a metastatic site) from procedure performed =< 5 years prior to pre-registration must be available to submit for Central Laboratory review prior to registration

    * Exception: If there is no medically safe site for biopsy, Study Chair (Dr. Haddad) may waive this requirement
* REGISTRATION INCLUSION CRITERIA
* Registration must be completed =< 28 days of pre-registration
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Histological confirmation of HER2-expression (immunohistochemistry [IHC] 1-3+) on pre-registration biopsy. (HER2+ is defined by 2018 American Society of Clinical Oncology/College of American Pathologists [ASCO/CAP] guidelines)

  * NOTE: If pre-registration biopsy is HER2- by ASCO/CAP guidelines then both of the following must be true:

    * The patient's most recent prior biopsy (prior to the pre-registration biopsy) must be HER2+, AND
    * The managing provider must be planning to treat the patient with anti-HER2 therapy
* For Cohort B only: Histologic confirmation of ERalpha positive disease (>= 1% expression)
* Hemoglobin >= 9.0 g/dL (obtained =< 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 100,000/mm^3 (obtained =< 14 days prior to registration)
* Direct bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 14 days prior to registration)
* Aspartate transaminase (AST) =< 3 x ULN (=< 5 x ULN for patients with liver involvement) (obtained =< 14 days prior to registration)
* Calculated creatinine clearance >= 45 ml/min using the Cockcroft-Gault formula (obtained =< 14 days prior to registration)
* Cardiac ejection fraction (left ventricular ejection fraction [LVEF]) >= 50% by echocardiogram =< 28 days prior to registration
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Negative urine pregnancy test done =< 7 days prior to registration, for women of childbearing potential only

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Patient and his/her partner agree to use adequate contraception after providing written informed consent through 3 months after the last dose of TVB-2640, as follows:

  * For women: Compliant with a medically-approved contraceptive regimen during and for 3 months after the treatment period or documented to be surgically sterile or postmenopausal
  * For men: Compliant with a medically-approved contraceptive regimen during and for 3 months after the treatment period or documented to be surgically sterile; men whose sexual partners are of child-bearing potential must agree to use 2 methods of contraception prior to study entry, during the study, and for 3 months after the treatment period
* Willingness to provide mandatory tumor tissue and/or blood specimens for correlative research

Exclusion Criteria:

* PRE-REGISTRATION EXCLUSION CRITERIA
* Patients who previously discontinued trastuzumab due to unacceptable cardiac toxicity
* Patients with a history of LVEF decline to below 50% during or after prior trastuzumab or other HER2 directed therapy =< 6 months prior to pre-registration
* Patients with any class of New York Heart Association (NYHA) congestive heart failure (CHF) or heart failure with preserved ejection fraction (HFPEF)
* Patients with a history of known coronary artery disease or a myocardial infarction within 12 months prior to pre-registration
* Patients with persistently uncontrolled hypertension (systolic blood pressure [BP] > 160 mm Hg or diastolic BP > 100 mm Hg) despite optimal medical therapy
* Patients with known unstable angina pectoris
* Patients with a known history of serious cardiac arrhythmias requiring treatment (exception: controlled atrial fibrillation, paroxysmal supraventricular tachycardia)
* Patients with a prolonged corrected QT interval (QTc) interval (>= 450 ms)
* Leptomeningeal disease or uncontrolled brain metastasis

  * NOTE: Metastases treated by surgery and/or radiotherapy such that patient is neurologically stable and off steroids >= 4 weeks prior to preregistration are eligible
* Failure to recover from acute, reversible effects of prior therapy regardless of interval since last treatment

  * EXCEPTION: Grade 1 peripheral (sensory) neuropathy that has been stable for at least 3 months since completion of prior treatment
* Tumors involving spinal cord or heart
* Visceral crisis or lymphangitic spread

  * NOTE: Visceral crisis is not the mere presence of visceral metastases, but implies severe organ dysfunction as assessed by symptoms and signs, laboratory studies, and rapid progression of disease
* Uncontrolled intercurrent non-cardiac illness including, but not limited to,

  * Ongoing or active infection
  * Psychiatric illness/social situations
  * Dyspnea at rest due to complications of advanced malignancy or other disease that requires continuous oxygen therapy
  * Or any other conditions that would limit compliance with study requirements
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Prior history of hypersensitivity, drug or radiation-induced, or other immune-mediated pneumonitis
* Patient is unable to swallow oral medications or has impairment of gastrointestinal (GI) function or GI disease that may significantly alter drug absorption (e.g. active inflammatory bowel disease, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome); note: concomitant therapy with proton pump inhibitors and/or H2-receptor antagonists is permissible
* Patient has a history of clinically significant dry eye (xerophthalmia) or other corneal abnormality, or if a contact lens wearer, does not agree to abstain from contact lens use from baseline through the last TVB-2640 dose
* Patients with a history of intolerance to trastuzumab (i.e. a grade 3 or 4 infusion reaction) are excluded; Note: patients with a history of mild infusion reaction to trastuzumab who have previously been successfully re-challenged after an infusion reaction with or without prophylactic medication are allowed
* Other invasive malignancy =< 3 years prior to pre-registration

  * EXCEPTIONS: Non-melanoma skin cancer, papillary thyroid cancer, or carcinoma-in-situ of the cervix which has been adequately treated
  * NOTE: If there is a history of prior malignancy, patients must not be receiving other treatment for their cancer and the disease must be inactive/stable
* REGISTRATION EXCLUSION CRITERIA
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Any of the following therapies prior to registration:

  * Chemotherapy =< 3 weeks
  * Immunotherapy =< 3 weeks
  * Biologic therapy =< 3 weeks
  * Monoclonal antibodies =< 3 weeks
  * Radiation therapy =< 2 weeks
  * CDK 4/6 inhibitors =< 4 weeks
  * mTOR inhibitors =< 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Up to 3 years
  Will be defined as the number of patients whose disease meets the Response Evaluation Criteria in Solid Tumors criteria for a partial or complete response on two consecutive evaluations at least 8 weeks apart divided by the total number of patients in that cohort who started protocol treatment. For each cohort, a two-stage Simon minimax design with a safety run-in period will be used to test the null hypothesis that the true tumor response rate is at most 5% against the alternative it is at least 20%.

SECONDARY OUTCOMES:
Duration of response | Up to 3 years
  Will be defined as the time from the first radiologic finding of a partial response or complete response to disease progression among those patients whose disease meets the Response Evaluation Criteria in Solid Tumors criteria for complete response or partial response on 2 consecutive evaluations approximately 8 weeks apart. A point and interval estimate of the response rate as well as the clinical benefit rate will be constructed using the Duffy-Santner approach to take into account the sequential nature of the study design. The distribution of response times and progression-free survival times will be estimated using the Kaplan-Meier approach.
Clinical benefit rate | Up to 3 years
  Will be defined as the proportion of patients who have completed 6 cycles of treatment without disease progression (that is, their objective disease status is a complete response, partial response, or stable for 6 cycles or more). A point and interval estimate of the response rate as well as the clinical benefit rate will be constructed using the Duffy-Santner approach to take into account the sequential nature of the study design. The distribution of response times and progression-free survival times will be estimated using the Kaplan-Meier approach.
Progression free survival | Up to 3 years
  Will be defined as time from randomization to the first of these disease events: local/regional or distant breast recurrence, ductal breast carcinoma in situ or invasive breast disease in contralateral breast, non-breast second primary, or death due to any cause. A point and interval estimate of the response rate as well as the clinical benefit rate will be constructed using the Duffy-Santner approach to take into account the sequential nature of the study design. The distribution of response times and progression-free survival times will be estimated using the Kaplan-Meier approach.

OTHER OUTCOMES:
Changes in biomarker expression | Baseline up to 28 days
  The changes in H score FASN, pAKT, and pS6 expression and levels of cellular apoptosis in tumor tissue will be examined graphically by plotting the difference in pre and post levels against pre-levels of the biomarker, with patients who derived clinical benefit represented by dashed line and those who did not by solid line. For each patient cohort, Wilcoxon signed rank tests will be used to assess the changes in serum FASN.

CONTACTS AND LOCATIONS:
Overall Officials: Tufia C. Haddad, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT03179904/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT03179904/ICF_001.pdf